CLINICAL TRIAL: NCT02189278
Title: Improving Adherence to Recommended Surveillance in Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00022895; 5K07CA138767 (NIH)
Record Dates: First submitted 2014-07-10; First posted 2014-07-14 (Estimated); Last update posted 2018-10-03 (Actual); Status verified 2018-09

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Surveillance; Mammography; Adherence
MeSH Terms: conditions — Breast Neoplasms | interventions — Psychosocial Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Psychosocial Intervention (Experimental): Telephone-based psychosocial intervention involving six telephone encounters. Each encounter focuses on teaching skills for improving adherence and overcoming barriers to obtaining recommended surveillance.
  Interventions: Behavioral: Psychosocial Intervention
- Treatment as usual (No Intervention): Treatment as usual control.

INTERVENTIONS:
Behavioral: Psychosocial Intervention — Telephone-based psychosocial intervention involving six telephone encounters. Each encounter focuses on teaching skills for improving adherence and overcoming barriers to obtaining recommended surveillance.
  Arms: Psychosocial Intervention

SUMMARY:
Evidence-based guidelines recommend cancer surveillance procedures for breast cancer survivors including physical examination, mammography, breast self-exam, and gynecologic follow-up. The early detection of recurrent and new cancers can best be achieved through the combined, on schedule use of these surveillance procedures. Yet, data suggest that up to 55% of breast cancer survivors do not undergo these procedures as recommended. This study tests a telephone-based psychosocial intervention aimed at improving adherence to recommended surveillance in breast cancer survivors. The psychosocial intervention for improving adherence is compared to treatment as usual.

ELIGIBILITY:
Inclusion Criteria:

* 21 years of age or older
* Diagnosis of Stage I to IIIA breast cancer
* Within 1 to 5 years post primary cancer treatment (i.e., surgery, chemotherapy, and/or radiation therapy)
* No diagnosis of recurrent breast cancer or a new primary cancer
* Able to provide meaningful consent

Exclusion Criteria:

* < 21 years of age
* Unable to provide meaningful consent
* Surgically treated with bilateral mastectomy

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-10; Primary Completion 2017-06-12 (Actual); Study Completion 2017-06-12 (Actual)

PRIMARY OUTCOMES:
Surveillance adherence | 15 month follow-up
  Receipt of recommended mammograms and clinical breast exams (coded 0=no, 1=yes)

SECONDARY OUTCOMES:
Gynecologic exam adherence | 15 month follow-up
  Receipt of recommended gynecologic exams (coded 0=no, 1=yes)
Breast self-exam adherence | 6 month follow-up
  Frequency of conducting breast self-exams assessed via patient report.

OTHER OUTCOMES:
Perceived benefits of surveillance | 6 month follow-up
  Patient reported perceived benefits of breast cancer surveillance
Perceived barriers to breast cancer surveillance | 6 month follow-up
  Patient reported perceived barriers to completing recommended breast cancer surveillance

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca A Shelby, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States